CLINICAL TRIAL: NCT05516472
Title: Fecal Microbiota Transplantation (FMT CAPSULE DE, FMPCapDE, MTP-CP101) in Kidney Stone Patients (FMT IND STUDY)
Brief Title: Fecal Microbiota Transplantation in Kidney Stone Patients
Acronym: FMT IND
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Joshua Stern (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor-Investigator, Joshua Stern, Chief of Urology, Intermountain Health Care, Inc.
Organization: Intermountain Health Care, Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1051917
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Kidney Stones
Keywords: microbial transplant therapy; kidney stones
MeSH Terms: conditions — Kidney Calculi | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, placebo-controlled
Who Masked: Participant
Masking Description: single-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Hyperoxaluric group (Experimental): Treatment group based on 24 hour urine analysis showing oxalate >40 mg/day.
  Interventions: Drug: Microbial Transplant Therapy
- Hypercalciuric Group (Experimental): Treatment group based on 24 hour urine analysis showing urinary calcium >225 mg/day.
  Interventions: Drug: Microbial Transplant Therapy
- Control group Hyperoxaluria (Placebo Comparator): Control group enrolling patients with hyperoxaluria
  Interventions: Drug: Placebo
- Control group Hypercalciuria (Placebo Comparator): Control group enrolling patients with hypercalciuria
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Microbial Transplant Therapy — Participants will take microbial capsules, 2 capsules daily for 7 days
  Other Names: fecal transplant
  Arms: Hypercalciuric Group; Hyperoxaluric group
Drug: Placebo — Participants will take placebo capsules
  Arms: Control group Hypercalciuria; Control group Hyperoxaluria

SUMMARY:
The purpose of this study is to measure the impact of Microbial Transplant Therapy (MTT) on 24-hour urine parameters in recurrent hypercalciuric and hyperoxaluric kidney stone formers.

DETAILED DESCRIPTION:
In this study, urinary stone disease patients will be recruited from the Park City Urology Clinic at Intermountain Healthcare.

Subjects will undergo screening and baseline assessments, including a history and physical exam. A 24-hour urine sample will be collected. Urinary parameters include analysis for calcium, oxalate, uric acid, citrate, NH4, sulfate, pH, Cr, phosphate, sodium, potassium, magnesium, super saturation (SS) CaOx, SSUA, SSCaP, UUN.

Microbial Transplant Therapy (MTT), the intervention, will be offered to individuals who produce greater than or equal to 50% calcium-oxalate stones. Pathology reports in the patient's medical record will be used to confirm the stone composition. The cohort of 36 total enrollees will be comprised of four separate study groups. The first group of 12 will include hyperoxaluric patients, the second group of 12 will include hypercalciuric patients, the third group will enroll six patients with hyperoxaluria as a control group, and the fourth group will enroll six patients with hypercalciuria as a control group. Grouping will be determined by 24-hour urine analysis which show measurements of urinary calcium greater than 225mg/day (hypercalciuric group) and oxalate greater than 40mg/day (hyperoxaluric group).

Stool samples will be obtained for metagenomic analyses prior to the intervention.

The study will begin with a run- in of 7 - 10 treatment patients, which will be followed by the randomization period.

In the randomization period, subjects will be assigned to the hypercalciuric and hyperoxaluric arms based upon urine parameters or placed in the control arm by random assignment. Because antibiotic treatment is common during surgery for stones, participants will be treated with 3 days of vancomycin 500 mg orally twice a day and neomycin 1,000 mg orally twice a day. This treatment is for all subjects, rather than only for subjects with recent or planned urological intervention; in order for the MTT to take hold, all patients must be treated with antibiotics. Forty-eight to 72 hours later, participants will take either the control capsule or the microbial capsules, 2 capsules daily for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Women and men age greater than or equal to 18 and less than 70
* Recent medical history of USD with greater than or equal to 50% calcium-oxalate stones. All patients will have urinary stone disease confirmed by stone analysis. The study will include patients with either stones extracted by urological intervention or spontaneously passed and collected stones.
* 24-hour urinary calcium concentration greater than 225 mg/day or urinary oxalate greater than 40 mg/day
* Able to give informed consent.
* Willing to undergo telephone follow-up to assess for safety and adverse events
* Willing and able to participate in the study requirements, including study visits, 24-hour urine collection and serial stool collection
* Not actively participating in another interventional USD clinical trial
* Estimated Glomerular Filtration Rate (eGFR) greater than or equal to 60.

Exclusion Criteria:

* Presence of three features of metabolic syndrome as defined by the NIH to have 3 or more of the following conditions:

  * Large waist - A waistline that measures at least 35 inches (89 centimeters) for women and 40 inches (102 centimeters) for men
  * High triglyceride level - 150 milligrams per deciliter (mg/dL), or 1.7 millimoles per liter (mmol/L), or higher of this type of fat found in blood
  * Reduced good or HDL cholesterol - Less than 40 mg/dL (1.04 mmol/L) in men or less than 50 mg/dL (1.3 mmol/L) in women of high-density lipoprotein (HDL) cholesterol
  * Increased blood pressure - 130/85 millimeters of mercury (mm Hg) or higher
  * Elevated fasting blood sugar - 100 mg/dL (5.6 mmol/L) or higher
* Presence of features of autoimmunity
* Major gastrointestinal surgery (e.g. significant bowel resection) within 3 months before enrollment. This does not include appendectomy or cholecystectomy
* Diagnosis of inflammatory bowel disease
* Patient diagnosed with primary hyperparathyroidism. Any patient with a PTH outside the range of 15 - 65 pg/ml will be excluded.
* Patient diagnosed secondary hyperparathyroidism. Any patient with a PTH outside the range of 15 - 65 pg/ml will be excluded.
* All patients requiring pancreatic enzyme replacement will be excluded.
* Patient with ongoing dialysis treatment
* Received chemotherapy treatment in the last 1 year
* Treatment with antibiotics within 3 months of study entry. If subjects need to take antibiotics unexpectedly during the trial, they are excluded if they have already taken the fecal material transplant; if not, they can re-enroll in 3 months.
* Patients taking potassium citrate, thiazides, or proton pump inhibitors in the last 6 months
* Women who are pregnant or breast-feeding or planning to get pregnant during the time of the study.
* Inability (e.g. dysphagia) to or unwilling to swallow capsules. Subjects with Grade greater than or equal to 2 dysphagia- as per Current Terminology for Common Adverse Events (CTCAE v 5.0) will be excluded.
* Active gastrointestinal infection at time of enrollment
* Requires continued antibiotic use or anticipates antibiotic use in the upcoming 4 weeks
* Known or suspected toxic megacolon and/or known small bowel ileus
* History of total colectomy or bariatric surgery
* Concurrent intensive induction chemotherapy, radiation therapy or biological treatment for active malignancy
* Expected life expectancy less than 6 months
* Previous FMT or microbiome-based products at any time excluding this study
* Patients with a history of severe anaphylactic or anaphylactoid food allergy
* Solid organ transplant recipients (all patients with a history of solid organ transplant will be excluded).
* A condition that would jeopardize the safety or rights of the subject, would make it unlikely for the subject to complete the study, or would confound the results of the study.
* Subjects will be excluded if they have chronic kidney disease defined as GFR (Glomerular Filtration Rate) less than 60.
* Subjects with urinary oxalate greater than or equal to 80 mg/d will be excluded

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with an adverse event | Baseline to day 30 (plus or minus 3 days) after fecal transplant
Changes in 24 hour urinary oxalate concentration | Baseline to weeks 1, 3, and 5
Changes in 24 hour urinary calcium concentration | Baseline to week 1, 3, and 5

SECONDARY OUTCOMES:
Metagenomic changes to subject microbiota pre-MTT | Prior to fecal transplant (baseline)
Metagenomic changes to subject microbiota post-MTT | weeks 4 and 5 after MTT

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Stern, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Park City Hospital, Park City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
The results of this study will be shared with the external collaborators on this study as per the clinical research agreement and as defined in the informed consent document.
Supporting Information: Study Protocol